CLINICAL TRIAL: NCT00309283
Title: Effect of a Long-acting Somatostatin on Disease Progression in Nephropathy Due to Autosomal Dominant Polycystic Kidney Disease: a Long-term Three Year Follow up Study
Brief Title: Somatostatin in Polycystic Kidney: a Long-term Three Year Follow up Study
Acronym: ALADIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALADIN; 2005-005552-41 (EudraCT Number)
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- somatostatin (Experimental)
  Interventions: Drug: Long-acting somatostatin
- Saline solution (Placebo Comparator)
  Interventions: Other: Saline solution

INTERVENTIONS:
Drug: Long-acting somatostatin — Patients randomized to treatment will be given intramuscularly long-acting somatostatin (Sandostatin-LAR, Novartis, Basel) at the dose of 40 mg every 28 days (in two intragluteal 20 mg injections).
  Arms: somatostatin
Other: Saline solution — Patients randomized to placebo will be given intramuscularly the same volume of solvent used to dissolve somatostatin every 28 days (in two intragluteal injections).
  Arms: Saline solution

SUMMARY:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) is the most common hereditary renal disease, responsible for 8% to 10% of the cases of end stage renal disease (ESRD) in Western countries. At comparable levels of blood pressure control and proteinuria, patients with ADPKD have faster decline in glomerular filtration rate than those with other renal diseases and do not seem to benefit to the same extent of ACE inhibitor therapy. A reasonable explanation for the above findings is that in ADPKD progression is largely dependent on the development and growth of cysts and secondary disruption of normal tissue. Thus, renoprotective interventions in ADPKD - in addition to achieve maximal reduction of arterial blood pressure and proteinuria and to limit the effects of additional potential promoters of disease progression such as dyslipidemia, chronic hyperglycemia or smoking - should also be specifically aimed to correct the dysregulation of epithelial cell growth, secretion, and matrix interactions characteristic of the disease.

Evidence that specific receptors for somatostatin are present in the kidney tissue, arises the possibility that somatostatin treatment in patients with ADPKD might inhibit fluid formation and eventually induce the shrinking of renal cysts.To evaluate the tolerability and the safety of long-acting somatostatin in ADPKD patients, a prospective cross-over controlled study has been recently performed. This pilot study demonstrated the safety of six month treatment of long-acting somatostatin in patients with ADPKD. Moreover, the percent increase of total kidney volume was significantly lower in patients on somatostatin than in placebo. Overall, these findings provide the basis for designing a long-term study in ADPKD patients aimed to document the efficacy of the somatostatin treatment in preventing further increase or even reducing the total kidney volume and the renal volume taken up by small cysts, eventually halting kidney disease progression.

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) is the most common hereditary renal disease, responsible for 8% to 10% of the cases of end stage renal disease (ESRD) in Western countries.

At comparable levels of blood pressure control and proteinuria, patients with ADPKD have faster decline in glomerular filtration rate (GFR) than those with other renal diseases and do not seem to benefit to the same extent of ACE inhibitor therapy. A reasonable explanation for the above findings is that in ADPKD progression is largely dependent on the development and growth of cysts and secondary disruption of normal tissue. Thus, renoprotective interventions in ADPKD - in addition to achieve maximal reduction of arterial blood pressure and proteinuria and to limit the effects of additional potential promoters of disease progression such as dyslipidemia, chronic hyperglycemia or smoking - should also be specifically aimed to correct the dysregulation of epithelial cell growth, secretion, and matrix interactions characteristic of the disease.

The fluid filling renal cysts in human polycystic kidney is formed mainly by a secretion process of the tubular epithelium lining the cysts. Secretion and re-absorption take place at approximately the same rate, with secretion slightly higher, so that the amount of fluid in the cysts increases slowly over time. The same process, via the secondary active chloride transport, is also involved in the secretion of fluid into the lumen of proximal tubules in teleost and elasmobranch fishes. Of interest, this process of chloride transport can be markedly inhibited by somatostatin, as demonstrated in the shark rectal gland.

Recently, somatostatin analogues have become available and used with negligible side effects for long-term treatment of tumors (up to 8-12 months). To evaluate the tolerability and the safety of long-acting somatostatin in ADPKD patients, a prospective cross-over controlled study has been recently performed. This pilot study demonstrated the safety of six month treatment of long-acting somatostatin in patients with ADPKD. Moreover, the percent increase of total kidney volume was significantly lower in patients on somatostatin than in placebo. Preliminary data on late stage ADPKD also suggest that loss of renal function in these patients closely correlates with the increase in kidney volume taken by small cysts (<5 mm3), but not total cyst volume.

Overall, these findings provide the basis for designing a long-term study in ADPKD patients aimed to document the efficacy of the somatostatin treatment in preventing further increase or even reducing the total kidney volume and the renal volume taken up by small cysts, eventually halting kidney disease progression.

Aims

The general aim of the study is to compare the effects on disease progression of three year treatment with long-acting somatostatin or placebo in patients with ADPKD and normal renal function or mild to moderate renal insufficiency. Specifically, the following aims will be pursued:

Primary To compare in somatostatin and placebo ADPKD groups the change over baseline of the total kidney volume at 1 and 3 years follow-up (estimated by gadolinium contrast enhanced and T2-weighted magnetic resonance imaging, MRI).

Secondary

1. As secondary efficacy endpoints, the following parameters (absolute and percent change over baseline by MRI analysis) will be compared in the two ADPKD groups at baseline, at 1 and 3 years follow-up:

   * Renal cyst volume
   * Total renal parenchymal volume
   * Residual renal volume
   * Renal parenchymal volume taken up by small cysts (<5 mm3)
2. Additional functional parameters will be compared in the two groups at baseline and at 1, 2, 3 years follow-up as follows:

   * Systolic and diastolic blood pressure
   * GFR (plasma iohexol clearance)
   * GFR (over baseline)
   * RPF (plasma PAH clearance)
   * Serum creatinine concentration
   * Diuresis
   * 24 h urinary protein excretion rate
   * 24 h urinary albumin excretion rate
   * Protein, albumin, creatinine concentrations on spot morning urine samples
   * Protein /creatinine ratio on spot morning urine samples
   * Albumin/creatinine ratio on spot morning urine samples
   * Urinary sodium, urea, glucose, phosphorus concentrations (24 hr samples)
   * Urine osmolality (calculated)
3. Correlation analyses between MRI and functional parameters will be also performed

Patients Patients enrolled in this long-term follow-up study are those with ADPKD and normal renal function or mild to moderate renal insufficiency (estimated GFR >40 ml/min/1.73 m2 by MDRD equation), no evidence of associated systemic, renal parenchymal or urinary tract disease and no specific contraindication to the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Clinical and ultrasound diagnosis of ADPKD
* GFR >40 ml/min/1-73 m2 (estimated by the 4 variable MDRD equation)
* Written informed consent

Exclusion Criteria

* Diabetes
* Overt proteinuria (urinary protein excretion rate >1g/24 hours) or abnormal urinalysis suggestive of concomitant, clinically significant glomerular disease
* Urinary tract lithiasis, infection or obstruction
* Cancer
* Psychiatric disorders and any condition that might prevent full comprehension of the purposes and risks of the study
* Pregnancy, lactation or child bearing potential and ineffective contraception (estrogen therapy in post menopausal women should not be stopped)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change over baseline of the total kidney volume at 1 and 3 years follow-up (estimated by gadolinium contrast enhanced and T2-weighted magnetic resonance imaging, MRI). | Basal, 1 and 3 years follow-up

SECONDARY OUTCOMES:
Absolute and percent change over baseline by MRI analysis will be compared in the two ADPKD groups at baseline, at one and three years follow-up of: | Basal, 1 and 3 years follow-up
Total renal parenchymal volume | Basal, 1 and 3 years follow-up
Residual renal volume | Basal, 1 and 3 years follow-up
Renal parenchymal volume taken up by small cysts, minor of five mmcubic | Basal, 1 and 3 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Perico, MD, Principal Investigator — Mario Negri Institute for Pharmacological Research
Locations (5):
- Italy (5):
  - University "Federico II" of Naples, Napoli, Napoli
  - Hospital Cà Foncello, Treviso, Treviso
  - Hospital "Ospedali Riuniti" Unit of Nephrology and Dialysis, Bergamo
  - Hospital "V. Fazzi" - Unit of neprology and Dialysis, Lecce
  - Hospital "Presidio Osp. Maggiore Policlinico", Milan

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Caroli A, Perico N, Perna A, Antiga L, Brambilla P, Pisani A, Visciano B, Imbriaco M, Messa P, Cerutti R, Dugo M, Cancian L, Buongiorno E, De Pascalis A, Gaspari F, Carrara F, Rubis N, Prandini S, Remuzzi A, Remuzzi G, Ruggenenti P; ALADIN study group. Effect of longacting somatostatin analogue on kidney and cyst growth in autosomal dominant polycystic kidney disease (ALADIN): a randomised, placebo-controlled, multicentre trial. Lancet. 2013 Nov 2;382(9903):1485-95. doi: 10.1016/S0140-6736(13)61407-5. Epub 2013 Aug 21. PMID 23972263